CLINICAL TRIAL: NCT04408742
Title: The Relationship Between Pain, Anxiety and Fatigue and Knee Position Sense, Balance and Dual Task Performance During Menstrual Cycle in Females With Multiple Sclerosis
Brief Title: Relationship Between Pain, Anxiety and Fatigue and Knee Position Sense, Balance and Dual Task Performance During Menstrual Cycle in Females With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019
Record Dates: First submitted 2020-05-26; First posted 2020-05-29 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Multiple Sclerosis; Menstrual Pain; Anxiety; Fatigue; Neurologic Symptoms
Keywords: multiple Sclerosis; menstrual cycle; proprioception; postural balance; pain; fatigue; anxiety
MeSH Terms: conditions — Multiple Sclerosis; Dysmenorrhea; Anxiety Disorders; Fatigue; Neurologic Manifestations; Pain | interventions — Proprioception

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- females with Multiple Sclerosis: patients with a confirmed diagnosis of MS according to the McDonald criteria, physician-administered Expanded Disability Status Scale (EDSS) range of 1-3.5, having regular menstrual cycle (between 21-35 days), and cognitive levels to give history and following the instructions
  Interventions: Other: pain; Other: fatigue; Other: anxiety; Other: position sense; Other: balance; Other: dual task performance

INTERVENTIONS:
Other: pain — Lower abdominal and low back pain was questioned. Pain intensity was evaluated with a 0 to 10 cm visual analog scale (VAS): "0" indicated "no pain" and "10" indicated "the worst imaginable pain [18]. Pain that developed during the activity was also questioned and stated as pain+ activity. A higher score indicates a more severe pain.
Other: fatigue — Fatigue was assessed by the Fatigue Severity Scale (FSS). This is a 9-item questionnaire that assesses the effect of fatigue on daily living. Each item is a statement on fatigue that the subject rates from 1 "completely disagree" to 7 "completely agree". A score of 4 or higher generally indicates severe fatigue.
Other: anxiety — The Spielberger State Trait Anxiety Inventory (STAI) was used to evaluate levels of anxiety. The state part of the STAI is a 20-item self-report inventory designed to measure state anxiety (current feelings of apprehension, worry, etc.). The STAI state scale is scored on four levels of anxiety intensity from 1 "not at all" to 4 "very much" and with a total score between 20 and 80. A higher total score indicates a more severe anxiety level.
Other: position sense — Knee position sense was evaluated with a Acumar dual digital inclinometer. Each participant was asked to wear shorts and to lie down in supine position treatment table. The lower extremity of the participant was positioned in neutral for the knee flexion movement. The placement of the digital inclinometer's attachment was the lateral ridge of the femur and tibia. We actively assisted the participant's knee to the target angle and asked the participant to hold it there for 5 seconds before returning the knee to the starting position. After returning to the starting position, participants attempted to repeat the previously attained angle. Participants indicated verbally when they felt they had reached the angle and held their position. This procedure was repeated 3 times for each limb (non-dominant and dominant). We measured the absolute difference between the target angle and the observed angle and calculated the absolute error score by averaging the 3 trials.
Other: balance — The Biodex Balance System (Biodex Medical Systems, Shirley, NY, USA) was used to measure limits of stability. The participants were asked to position themselves in a comfortable position on the platform and their foot position coordinate was recorded. The participants were asked to complete as quickly as possible the directional tasks displayed on a screen, with the directions displayed at random. A total of 3 tests were performed, at intervals of 10 s. A total score was recorded. The higher the total score, the better the ability of the subjects to transfer the center of gravity.
Other: dual task performance — The timed up and go test (TUG) was used in the evaluation of dual task performance. For this test, participants were seated on a standard armless chair and a cone was placed 3 meters away from the chair. Participants were instructed to stand up and (1) walk towards the cone, (2) turn around the cone, (3) walk back to the chair, and (4) sit back on the chair. It was stated that patients should walk without running but as fast as possible. TUG test was performed initially without task, and then with cognitive and motor tasks, respectively. Cognitive task given during the test is counting three backwards from 100 or counting the names starting with the letter "A", and motor task given is to carry three glasses of water on a tray. The time elapses between standing up from the chair and sitting back to chair was recorded as the test result. As time increases, dual task performance decreases.

SUMMARY:
This study was carried out to investigate the relationship between pain, anxiety and fatigue and knee position sense, balance and dual task performance during menstrual cycle in females with Multiple Sclerosis (FwMS).

In the neurologic group, especially in MS patients, it is well known that disease activity, course, and symptoms can be influenced by the menstrual cycle. Previous studies have reported that the fluctuations of estrogen and progesterone during the menstrual cycle may have an effect on several neurological functions. Menstrual-related symptomatology has primarily been studied as a physiological phenomenon. Increased neurological symptoms, physical disorders and behavioral changes have been reported just before or at the beginning of menstruation in FwMS.

For all these reasons,investigators think that relationship between pain, anxiety and fatigue and knee position sense, balance and dual task performance during menstrual cycle in FwMS.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria were as follows: patients with a confirmed diagnosis of MS according to the McDonald criteria, physician-administered Expanded Disability Status Scale (EDSS) range of 1-3.5, having regular menstrual cycle (between 21-35 days), and cognitive levels to give history and following the instructions.

Exclusion Criteria:

The exclusion criteria were: patients with acute attacks and using corticosteroid (three months prior to the study), taking oral contraceptive agents, and history of orthopedic lower extremity problems or other neurological disorders.

Ages: 26 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — having regular menstrual cycle females with MS
Study Population: patients with a confirmed diagnosis of clinically definite MS, physician-administered Expanded Disability Status Scale (EDSS) range of 1-3.5, and having regular menstrual cycle (between 21-35 days).
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-10-20 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
pain intensity | through study completion, an average of 1 year
  Pain intensity was evaluated with a 0 to 10 cm visual analog scale (VAS): "0" indicated "no pain" and "10" indicated "the worst imaginable pain. A higher score indicates a more severe pain.
anxiety | through study completion, an average of 1 year
  The Spielberger State Trait Anxiety Inventory was used to evaluate levels of anxiety.The state part of the STAI is a 20-item self-report inventory designed to measure state anxiety. A higher total score indicates a more severe anxiety level.
fatigue | through study completion, an average of 1 year
  Fatigue was assessed by the Fatigue Severity Scale. Each item is a statement on fatigue that the subject rates from 1 "completely disagree" to 7 "completely agree". A score of 4 or higher generally indicates severe fatigue.
position sense | through study completion, an average of 1 year
  Knee position sense was evaluated with a Acumar dual digital inclinometer.The absolute error scores (in degrees) for knee flexion at 60° was calculated. As absolute error score increases, position sense decreases.
balance | through study completion, an average of 1 year
  The participants are asked to complete the directional tasks displayed on a screen as quickly as possible, with the directions displayed at random. A total of 3 tests were performed, at intervals of 10 second. The test results were used to determine a total score. The higher the total score, the better the ability of the subjects to transfer the centre of gravity.
dual task performance | through study completion, an average of 1 year
  The timed up and go test was used in the evaluation of dual task performance. Timed up and go test was performed initially without task, and then with cognitive and motor tasks, respectively. Cognitive task given during the test is counting three backwards from 100 or counting the names starting with the letter "A", and motor task given is to carry three glasses of water on a tray. The time elapses between standing up from the chair and sitting back to chair was recorded as the test result. As time increases, dual task performance decreases.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences,Department of Physiotherapy and Rehabilitation, Ankara, Esenboğa, Turkey (Türkiye)

REFERENCES:
- [Derived] Ates Y, Unluer NO. The relationship of pain, anxiety, and fatigue with knee position sense, balance, and dual task performance during menstrual cycle in females with multiple sclerosis. Somatosens Mot Res. 2020 Dec;37(4):307-312. doi: 10.1080/08990220.2020.1828057. Epub 2020 Oct 7. PMID 33026291